CLINICAL TRIAL: NCT05200611
Title: Application of Fecal Immunochemical Test for Improving Advanced Adenoma Detection in Colorectal Cancer Screening
Brief Title: Fecal Immunochemical Test for Advanced Adenoma Detection in Colorectal Cancer Screening
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Collaborators: The People's Hospital of Zhaoyuan City (Unknown); Shanghe People's Hospital (Unknown)
Responsible Party: Principal Investigator, Yanqing Li, Clinical Professor, Shandong University
Other Study IDs: 2022SDU-QILU-103
Record Dates: First submitted 2022-01-03; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Colorectal Cancer; Colorectal Neoplasms; Colorectal Adenoma
Keywords: Colorectal Adenoma; Occult Bleeding; Quantitative fecal immunochemical test
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — faeces
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fecal Immunochemical Test: People in this group with positive fecal immunochemical test results were further examined by colonoscopy.
  Interventions: Diagnostic Test: Fecal Immunochemical Test

INTERVENTIONS:
Diagnostic Test: Fecal Immunochemical Test — Participants with positive fecal immunochemical test results were further examined by colonoscopy.

SUMMARY:
Early detecting and removing of colorectal advanced adenomas can reduce incidence of colorectal cancer. In order to reduce the incidence of colorectal cancer, improve the early diagnosis of colorectal cancer, the investigators conducted this study to explore diagnostic accuracy of fecal immunochemical test in colorectal cancer screening population.

DETAILED DESCRIPTION:
Colorectal cancer accounts for approximately 10% of all annually diagnosed cancers and cancer-related deaths worldwide. With progress of developing countries, it is predicted that the incidence of colorectal cancer worldwide will increase to 2.5 million new cases in 2035. The majority of colorectal cancer is thought to arise from precancerous lesions through the adenoma-carcinoma pathway. Detecting and removing of colorectal advanced adenomas can reduce incidence of colorectal cancer. In order to reduce the incidence of colorectal cancer, improve the early diagnosis of colorectal cancer, the investigators conducted this study to explore diagnostic accuracy of fecal immunochemical test in colorectal cancer screening population.

ELIGIBILITY:
Inclusion Criteria:

* Adults 50-75 years old

Exclusion Criteria:

* People with history of intestinal surgery;
* People with history of colorectal cancer;
* People with history of inflammatory bowel disease, ischemic enteritis, vascular malformation of intestine or other disease resulting in intestinal tract bleeding;
* People with symptoms including visible rectal bleeding, hematuria, severe and acute diarrhea;
* Pregnancy, lactation or menstrual phase;
* Severe congestive heart failure or other sever disease cause cannot tolerate colonoscopy.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Continuous participants intending to undergo colonoscopy and meet the inclusion and exclusion criteria were enrolled.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
The efficacy of fecal immunochemical test to detect advanced adenoma | 6 months
  The detection rate and positive predictive value of fecal immunochemical test to detect advanced adenoma

SECONDARY OUTCOMES:
The efficacy of fecal immunochemical test to detect colorectal cancer | 6 month
  The detection rate and positive predictive value of fecal immunochemical test to detect colorectal cancer
The efficacy of fecal immunochemical test to detect colorectal neoplasms | 6 month
  The detection rate and positive predictive value of fecal immunochemical test to detect colorectal neoplasms

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Shanghe People's Hospital, Jinan, Shandong
  - The People's Hospital of Zhaoyuan City, Yantai, Shandong